CLINICAL TRIAL: NCT00922948
Title: A Prospective Randomized Pilot Trial of Cryoablation (CA) Versus Radio Frequency Ablation (RFA) for the Management of Small Renal Masses
Brief Title: Cryoablation Versus Radiofrequency Ablation for Small Renal Masses
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cryoablation is no longer offered at our hospital, and likely won't be offered in the near future.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-001-09
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Renal Cancers
Keywords: Radiofrequency ablation; Cryosurgery; Renal cancers
MeSH Terms: conditions — Kidney Neoplasms | interventions — Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryoablation (Experimental)
  Interventions: Procedure: Cryoablation
- Radiofrequency ablation (Active Comparator): Radiofrequency ablation
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Cryoablation — Cryoneedles and one temperature probe are inserted under endoscopic and sonographic guidance.
  Arms: Cryoablation
Procedure: Radiofrequency ablation — Thermal injury is the predominant mechanism of action of RFA. A high-frequency alternating current emitted from the exposed noninsulated portion of the electrode generates frictional heat, agitating ions in the tissue surrounding the tip of the needle.
  Arms: Radiofrequency ablation

SUMMARY:
The purpose of this study is to verify the oncological efficacy and safety of cryoablation and radiofrequency ablation for the treatment of small renal tumors.

DETAILED DESCRIPTION:
By enrolling all patients treated with CA or RFA, this study will document for the first time the safety and the short and long term efficacy of CA compared to RFA as well as provide urologists and decision makers currently unavailable information on CA in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors that progress in size while on a watchful waiting protocol;
* Patients with multiple tumors;
* Patients with a tumor in a solitary kidney;
* Patients with poor renal function and a renal tumor;
* Patients with significant co-morbidities that may benefit from a less invasive approach.

Exclusion Criteria:

* Large tumors > 4.0cm;
* Unable to have a general anesthetic;
* Unable to comply with follow-up protocol (i.e., routine CT or MRI and a follow-up biopsy);
* Uncorrectable bleeding diathesis;
* Evidence of metastatic disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Treatment failure rate. | Baseline, Weeks 6, 12, 24, 36, 48

SECONDARY OUTCOMES:
Renal function - GFR of less than 60 ml per min per 1.73 m2. Serum creatinine and creatinine clearance. | Baseline, Weeks 6, 12, 24, 36 and 48
Average percentage decrease in tumor size. | Baseline, Weeks 6, 12, 24, 36 and 48
Intra and post-operative complications rates. | Weeks 6, 12, 24, 36 and 48
Quality of life data. | Baseline, Weeks 6, 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, Principal Investigator — McMaster Institute of Urology, McMaster University
Locations (1):
- McMaster Institute of Urology - St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada